CLINICAL TRIAL: NCT00583206
Title: Biochemical Pathways to Skeletal Muscle Atrophy in Human Sepsis
Brief Title: Muscle Atrophy in Sepsis
Status: Withdrawn | Type: Observational
Sponsor: Gregory A. Schmidt (Other)
Responsible Party: Sponsor-Investigator, Gregory A. Schmidt, Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 200706755
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Atrophy; Sepsis; Weakness
Keywords: sepsis; atrophy; muscle; weakness
MeSH Terms: conditions — Atrophy; Sepsis; Asthenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Muscle RNA; blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Severe sepsis will provoke signals leading to muscle atrophy and weakness. Electrical stimulation will reduce the impact of sepsis.

DETAILED DESCRIPTION:
Hypothesis 1: Severe sepsis will be associated with downregulation of anabolic signaling molecules and genes, upregulation of catabolic signaling molecules and genes, and the development of histologic and electrophysiologic abnormalities within skeletal muscle.

Hypothesis 2: Electrical stimulation will improve muscle strength in patients with sepsis.

Hypothesis 3: Electrical stimulation will be associated with upregulation of anabolic signaling molecules and genes, downregulation of catabolic signaling molecules and genes, and improvement of histologic and electrophysiologic parameters within skeletal muscle of patients with sepsis.

Hypothesis 4: The ratio of catabolic:anabolic gene expression on Day 3 will be positively correlated with the severity of clinical weakness on Day 7

ELIGIBILITY:
Inclusion Criteria:

* Severe sepsis for < 72hr

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe sepsis
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-12; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Electrical stimulation will be associated with upregulation of anabolic signaling molecules and genes, downregulation of catabolic signaling molecules and genes within skeletal muscle of patients with sepsis | 3 days

SECONDARY OUTCOMES:
Electrical stimulation will be associated with improvement of histologic and electrophysiologic and strength parameters within skeletal muscle of patients with sepsis | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Hospitals, Iowa City, Iowa, United States